CLINICAL TRIAL: NCT06951061
Title: Reproductive Outcomes in Children Born Through Assisted Reproduction (ART): Focus on Intracytoplasmic Sperm Injection (ICSI) With Surgically Retrieved Sperm.
Brief Title: Reproductive Outcomes After Intracytoplasmic Sperm Injection (ICSI) With Surgically Retrieved Sperm.
Acronym: SRS-ICSI outc
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Göteborg University (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Panagiotis Tsiartas, Associate Professor, Karolinska Institutet
Other Study IDs: 2025-00935-01
Record Dates: First submitted 2025-04-15; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Reproductive Technology, Assisted; IVF Outcomes; ICSI
Keywords: perinatal outcomes; IVF; ICSI; surgically retrieved sperm
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IVF with ejaculated sperm: This group have gone through IVF with ejaculated sperm. Both fresh and frozen cycles are included.
  Interventions: Procedure: IVF/ICSI
- ICSI with ejaculated sperm: This group have gone through ICSI with ejaculated sperm. Both fresh and frozen cycles are included.
  Interventions: Procedure: IVF/ICSI
- ICSI with surgically retrieved sperm: This group have gone through ICSI with surgically retrieved sperm. Both fresh and frozen cycles are included.
  Interventions: Procedure: IVF/ICSI

INTERVENTIONS:
Procedure: IVF/ICSI — In vitro fertilization with or without ICSI with ejaculated and surgically retrieved sperm.

SUMMARY:
This research project explores how the source of sperm affects outcomes in assisted reproductive technologies (ART), focusing on children conceived through intracytoplasmic sperm injection (ICSI) with surgically retrieved sperm (SRS). Outcomes will be compared to those from ICSI with ejaculated sperm and conventional IVF. Using national registry data from all IVF and ICSI treatments in Sweden between 2007 and 2023 (Q-IVF), the study applies artificial intelligence (AI) and machine learning (ML) to identify factors influencing success rates. The aim is to improve prediction models and support more personalized fertility treatments. Special emphasis is placed on understanding the potential risks and long-term health outcomes for children conceived using SRS, which may be associated with higher rates of genetic abnormalities. The results may help optimize care strategies for infertile couples.

DETAILED DESCRIPTION:
This research project aims to improve our understanding of how different sources of sperm affect outcomes in assisted reproductive technologies (ART). The focus is on children conceived through intracytoplasmic sperm injection (ICSI) using surgically retrieved sperm (SRS), compared to ICSI with ejaculated sperm and conventional in vitro fertilization (IVF).

The study has three main goals:

1. To compare reproductive outcomes following ICSI with SRS, ICSI with ejaculated sperm, and conventional IVF.
2. To investigate whether artificial intelligence (AI) and machine learning (ML) algorithms can predict cumulative reproductive outcomes, including results from both fresh and frozen embryo transfer cycles.
3. To evaluate how AI/ML-based models perform in comparison to traditional statistical methods in terms of accuracy and predictive value.

Method: National Population-Based Registry Study: This includes all IVF and ICSI treatments performed in Sweden from January 1, 2007, to December 31, 2023, using data from the Swedish National Quality Registry for Assisted Reproduction (Q-IVF). AI will be used to analyze large datasets, detect patterns, and help identify key factors-such as sperm source, number of retrieved oocytes, and patient characteristics-that may influence treatment success. This approach could lead to personalized treatment plans and better predictions of successful pregnancy outcomes.

Special attention is given to outcomes in children born after ICSI with surgically retrieved sperm, as these sperm may be less mature and carry a higher risk of genetic abnormalities. The findings are expected to provide valuable insights into the reproductive and long-term health outcomes of these treatments, ultimately helping to improve care and treatment strategies for infertile couples.

ELIGIBILITY:
Inclusion Criteria:

* All IVF treatments performed in Sweden during the study period.
* IVF treatments will be identified from the National register Q-IVF.

Exclusion Criteria:

* Children born from multiple pregnancies
* Children conceived through oocyte and sperm donation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In this population-based project, data from the National Quality Registry Q-IVF will be employed to identify a birth cohort comprising all IVF treatments performed in Sweden between January 1, 2007, and December 31, 2023. This time frame aligns with the establishment in 2007 of the National Quality Registry for Assisted Reproduction (Q-IVF). This cohort will be followed until December 31, 2023, resulting in a 16-year period.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical pregnancy rate | From enrollment to the end of treatment at 3 weeks
  Positive urinary pregnancy test after fresh or frozen embryo transfer per embryo transfer.
Clinical pregnancy rate | From enrollment to the end of treatment at 8 weeks.
  Presence of gestational sac at ultrasound control after fresh or frozen embryo transfer per embryo transfer.
Live birth rate | From enrollment to the end of treatment at delivery.
  Live birth per embryo transfer after fresh and frozen embryo transfer.

SECONDARY OUTCOMES:
Number of frozen embryos | From enrollment to the end of treatment at 5 days.
  Number of embryos at blastocyst stage that are frozen.
Miscarriage rate | From enrollment to the end of treatment before 22 weeks.
  Miscarriage per clinical pregnancy after fresh and frozen embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Tsiartas, Associate Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Clinical Science, Intervention and Technology, Division of Obstetrics and Gynaecology, Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the data will be retrieved from Q-IVF in anonymized form, ensuring that no individual can be identified. As such, there is no access to raw, identifiable data, and sharing is restricted to protect patient confidentiality and comply with data protection regulations.